CLINICAL TRIAL: NCT06834048
Title: Validity - Reliability of Berg Balance Scale in Albanian Population
Acronym: BERGA
Status: Recruiting | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jasemin Todri, Professor, Universidad Católica San Antonio de Murcia
Other Study IDs: 208
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Balance Assessment; Balance Control in Elderly; Balance Changes; Geriatric Assessment
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation alone — Psychometric properties will be assessed by administering the questionnaire online to approximately 200 participants. Reliability will be estimated by assessing stability and homogeneity.

SUMMARY:
Cross-cultural adaptation, validity and Reliability of Berg Balance Scale in Albanian population

DETAILED DESCRIPTION:
The cross-cultural adaptation will be carried out in accordance with the internationally recommended methodology, following the guidelines: translation, back-translation; dissemination of questionnaires and data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Postural pain
* muscular contractions

Exclusion Criteria:

* mixed fractures
* trauma
* luxation
* tumor

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: geriatric people with postural compensations
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Albanian Berg Balance Scale | 10 minutes
  This scale measures balance in older adults. It consist in 14 Items. Is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Jasemin Todri, Murcia, Spain